CLINICAL TRIAL: NCT05585450
Title: Effect of Electroacupuncture on Lower Urinary Tract Symptoms of Benign Prostatic Hyperplasia: a Randomized Controlled Trial
Brief Title: Effect of Electroacupuncture on Benign Prostatic Hyperplasia
Acronym: EABPH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Liu Zhishun, Chief Physician, Dean of Acupuncture Department, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-203-KY
Record Dates: First submitted 2022-10-13; First posted 2022-10-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: acupuncture; randomized controlled trial; lower urinary tract symptoms
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture (EA) group (Experimental): Participants in the EA group will receive treatment at bilateral Bladder Meridian (BL) 32 [Ciliao], BL33 [Zhongliao], BL35 [Huiyang], and Spleen Meridian (SP) 6 [Sanyinjiao].
  BL32, in the second posterior sacral foramen; BL33, in the third posterior sacral foramen; BL35, 0.5 cun (≈10mm) lateral to the extremity of the coccyx; SP6, posterior to the medial border of the tibia, 3 cun (≈60mm) superior to the prominence of the medial malleolus.
  The treatment will last 30 minutes for each session, 3 sessions per week (ideally every other day) for a succession of 8 weeks.
  Interventions: Device: Electroacupuncture
- Sham Electroacupuncture (SA) group (Sham Comparator): Participants in the SA group will receive treatment at bilateral sham BL32, BL33, BL35, and SP6.
  Sham BL32, in the area of 2 cun (≈40mm) horizontally outside BL32; Sham BL33, in the area of 2 cun (≈40mm) horizontally outside BL33; Sham BL35, 2 cun (≈40mm) horizontally outside BL35; Sham SP6, in the middle of SP6 and tendons.
  The treatment will last 30 minutes for each session, 3 sessions per week (ideally every other day) for a succession of 8 weeks.
  Interventions: Device: Sham electroacupuncture

INTERVENTIONS:
Device: Electroacupuncture — BL32 and BL33 will be inserted by needles of 0.30×75mm size at an angle of 45°, inward and downward, to the depth of 60-70mm. BL35 will be inserted by needles of 0.30×75mm size, slightly outward and upward, to the depth of 60-70mm. SP6 will be inserted by needles of 0.30×40mm to the depth of 25-30mm. The needles will be lifted, thrust, and twisted evenly three times after insertion to induce the sensation of deqi.
  The electronic acupuncture apparatus (Yingdi KWD 808I electro pulse acupuncture therapeutic apparatus, Changzhou Yingdi Electronic Medical Device Co., Ltd) will be connected to the four pairs of needles transversally, with a continuous wave of 5 Hertz (Hz) and an electric current of 2-6.5 milliampere (mA) for BL32, BL33 and BL35, and 0.5 mA-2mA for SP6.
  Other Names: EA
  Arms: Electroacupuncture (EA) group
Device: Sham electroacupuncture — The four pairs of acupoints will be inserted by needles of 0.30×25mm or 0.30×40mm size to a depth of 2-3mm till the needles can stand still. No manipulations will be conducted, and the sensation of deqi will not be induced.
  The electronic acupuncture apparatus (Yingdi KWD 808I electro pulse acupuncture therapeutic apparatus, Changzhou Yingdi Electronic Medical Device Co., Ltd) will be connected to the four pairs of needles transversally, with a continuous wave of 5 Hz and a minimal electric current (ideally at a degree which participant can just percept). In about 30 seconds, the electric current will be turned down, leaving the indicator light and ticking sound on.
  Other Names: SA
  Arms: Sham Electroacupuncture (SA) group

SUMMARY:
The study aims to assess the efficacy and safety of electroacupuncture among men with benign prostatic hyperplasia (BPH), compared with sham electroacupuncture.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of BPH in accordance with the European Association of Urology (EAU) guideline;
2. Male participants aged between 40 and 80 years;
3. Lower urinary tract symptoms (LUTS) for at least three months;
4. IPSS total score ≥8;
5. Prostate volume ≥20 mL;
6. Urinary peak flow rate (Qmax) ≤15 mL/s;
7. Voluntary participation in the trial and signed written informed content.

Exclusion Criteria:

1. Post-void residual urine volume (PVR) ≥150 mL;
2. Acute urinary retention or catheterization for outflow obstruction within the 3 months (Except for post-surgical disposable catheterization);
3. Prostate cancer or prostate-specific antigen (PSA) level ≥4.0 ng/mL;
4. Neurogenic lower urinary tract dysfunction; prostatitis; uncontrolled symptomatic urinary tract infections; urethral strictures; bladder diverticula; bladder stones; bladder cancer; history of genitourinary system surgery (prostate, bladder, urethra, etc.);
5. Previous acupuncture treatment for BPH in the preceding one month, or α-blockers, 5α-reductase inhibitor, muscarinic receptor antagonists, or any other specific medication usage in the previous two weeks unless a stable 5α-reductase inhibitor usage of over three months;
6. Severe lung, heart, liver, kidney, metabolic, or mental illness, coagulation dysfunction, or with obvious cognitive dysfunction;
7. Installed cardiac pacemaker, allergy to metal, severe fear of acupuncture or unbearable to the stimulation of EA.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants with at least 30% reduction in the total score of International Prostate Symptom Score (IPSS) from baseline | week 8
  The IPSS is a valid, reliable, and sensitive measure tool frequently used to evaluate the severity of lower urinary tract symptoms, including incomplete bladder emptying, frequency of urination, intermittency, urgency, weak urine stream, straining, and nocturia. The score of IPSS ranges from 0 to 35, with scores of 0 to 7 indicating mild symptoms; 8 to 19 indicating moderate symptoms; and 20 to 35 indicating severe symptoms.
The proportion of participants with at least 30% reduction in the total score of International Prostate Symptom Score (IPSS) from baseline | week 20
  The IPSS is a valid, reliable, and sensitive measure tool frequently used to evaluate the severity of lower urinary tract symptoms, including incomplete bladder emptying, frequency of urination, intermittency, urgency, weak urine stream, straining, and nocturia. The score of IPSS ranges from 0 to 35, with scores of 0 to 7 indicating mild symptoms; 8 to 19 indicating moderate symptoms; and 20 to 35 indicating severe symptoms.

SECONDARY OUTCOMES:
The change from baseline in the total score of IPSS | weeks 4, 8, 12, 20, 32
  The IPSS is a valid, reliable, and sensitive measure tool frequently used to evaluate the severity of lower urinary tract symptoms, including incomplete bladder emptying, frequency of urination, intermittency, urgency, weak urine stream, straining, and nocturia. The score of IPSS ranges from 0 to 35, with scores of 0 to 7 indicating mild symptoms; 8 to 19 indicating moderate symptoms; and 20 to 35 indicating severe symptoms.
The proportion of participants with at least 30% reduction in the total score of IPSS from baseline | weeks 4, 12, 32
  The IPSS is a valid, reliable, and sensitive measure tool frequently used to evaluate the severity of lower urinary tract symptoms, including incomplete bladder emptying, frequency of urination, intermittency, urgency, weak urine stream, straining, and nocturia. The score of IPSS ranges from 0 to 35, with scores of 0 to 7 indicating mild symptoms; 8 to 19 indicating moderate symptoms; and 20 to 35 indicating severe symptoms.
The proportion of participants with at least 50% reduction in the total score of IPSS from baseline | weeks 4, 8, 12, 20, 32
  The IPSS is a valid, reliable, and sensitive measure tool frequently used to evaluate the severity of lower urinary tract symptoms, including incomplete bladder emptying, frequency of urination, intermittency, urgency, weak urine stream, straining, and nocturia. The score of IPSS ranges from 0 to 35, with scores of 0 to 7 indicating mild symptoms; 8 to 19 indicating moderate symptoms; and 20 to 35 indicating severe symptoms.
The change from baseline in the voiding and storage subscale scores of IPSS | weeks 4, 8, 12, 20, 32
  The IPSS is a valid, reliable, and sensitive measure tool frequently used to evaluate the severity of lower urinary tract symptoms, including incomplete bladder emptying, frequency of urination, intermittency, urgency, weak urine stream, straining, and nocturia. The score of IPSS ranges from 0 to 35, with scores of 0 to 7 indicating mild symptoms; 8 to 19 indicating moderate symptoms; and 20 to 35 indicating severe symptoms.
The change from baseline in the number of nocturia | weeks 4, 8, 12, 20, 32
  Participants will be asked: During the last month, how many times did you most typically get up to urinate from the time you went to bed at night until the time you got up in the morning?
The change from baseline in the quality of life (QOL) item of IPSS | weeks 4, 8, 12, 20, 32
  Participants will be asked the question: If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that? The response categorized into 7 degrees scoring 0 to 6, respectively: 0 (delighted), 1 (pleased), 2 (mostly satisfied), 3 (mixed about equally satisfied and dissatisfied), 5 (mostly dissatisfied), 5 (unhappy), and 6 (terrible).
The change from baseline in the BPH Impact Index (BPH-II) | weeks 4, 8, 12, 20, 32
  The BPH-II measures the interference of LUTS in patients' mental health and activity. The total score of BPH-II ranges from 0 to 13, with higher scores indicating poorer quality of life.
The change from baseline in the International Index of Erectile Function 5 (IIEF-5) | weeks 8, 20, 32
  The IIEF-5 is a valid and reliable instrument for detecting treatment effects in patients with erection dysfunction, ranging from 1 to 25, with lower scores indicating more severe dysfunction.
The change from baseline in the hours of undisturbed sleep (HUS) | weeks 4, 8, 12, 20, 32
  HUS is defined as the duration from falling asleep till awake in the morning, or till the first nocturia if any.
The change from baseline in the Hospital Anxiety and Depression Scale (HADS) | weeks 8, 20, 32
  The HADS score ranges from 0 to 42, with higher scores indicating greater anxiety and depression.
The change from baseline in the volume of prostate | week 8
  The prostate volume will be measured by transabdominal ultrasound.
The change from baseline in the post-void residual urine volume | week 8
  The post-void residual urine volume will be measured by transabdominal ultrasound.
The change from baseline in the urinary peak and average flow rate | week 8
  The urinary peak and average flow rate will be measured by uroflowmetry.
The proportion of responders per the Patient Global Index of Improvement (PGI-I) | weeks 8, 20, 32
  The PGI-I evaluates the overall treatment effect perceived by patients themselves. The change can be rated in 7 levels, including "very much better", "much better", "a little better", "no change", "a little worse", "much worse" or "very much worse".

OTHER OUTCOMES:
Expectance assessment | Baseline assessment (week 0)
  Participants will be asked: How do you expect your lower urinary tract symptoms (LUTS) will be in two months?
Assessment of belief in acupuncture | Baseline assessment (week 0) and week 8
  Participants will be asked the question: Do you think your BPH may be helped by acupuncture? Time Frame: Baseline assessment (week 0) and week 8 Participants will be asked the question: Do you think your BPH may be helped by electroacupuncture?
Blinding assessment | Within 5 minutes after either treatment at week 8
  Participants will be asked the question: Do you think you have received traditional electroacupuncture in the past 8 weeks?
Safety assessment | Throughout the trial
  Adverse events and severe adverse events will be recorded in the case report form, whether related to interventions or not.
Adherence assessment | weeks 1-8
  Adherence will be assessed via counting treatment sessions. Those who complete over 80% treatment sessions will be defined as of good adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data and data dictionary will be available with the publication until six months after publication.
  A formal request should be sent to zhishunjournal@163.com with a methodologically sound proposal.
  Researchers whose proposal has been approved will sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available with the publication until six months after publication.
Access Criteria: A formal request should be sent to zhishunjournal@163.com with a methodologically sound proposal. Researchers whose proposal has been approved.
  Researchers whose proposal has been approved will sign a data access agreement.

REFERENCES:
- [Derived] Zhu L, Yan Y, Yu J, Liu Y, Sun Y, Chen Y, Fang J, Liu Z. Electroacupuncture for lower urinary tract symptoms in men with benign prostatic hyperplasia: study protocol for a randomised controlled trial. BMJ Open. 2024 Jul 20;14(7):e080743. doi: 10.1136/bmjopen-2023-080743. PMID 39032929